CLINICAL TRIAL: NCT03394495
Title: Evaluation of an Individualized Exercise Programme Plus Behavioural Change Enhancement Strategies for Managing General Fatigue in Community-dwelling Frail Older People: A Cluster-randomized Controlled Trial.
Brief Title: Individualized Exercise Program Plus Behavioral Change Enhancement Strategies for Managing Fatigue in Frail Older People
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Responsible Party: Principal Investigator, Dr. Justina Liu Yat Wa, Associate Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 15600717
Record Dates: First submitted 2017-12-15; First posted 2018-01-09 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Fatigue
Keywords: Fatigue; Frailty; Cluster-RCT; Exercise; Behavioral change
MeSH Terms: conditions — Fatigue; Frailty; Motor Activity

STUDY DESIGN:
Intervention Model Description: A three-arm parallel (single-blinded) cluster randomized controlled trial involves three groups of participants (the COMB, the EXER and the control group). Twelve community health centres that provide similar types of community care and social support services for community-dwelling older people, have been invited by a convenience method to work as collaborators in this study. Using computer-generated random numbers, a biostatistician not affiliated with this study will randomize the centres into either: control, EXER, or COMB group. So during the trial, participants in one group receive combination intervention "in parallel" to participants in the other two groups (the control group and the exercise group).
Who Masked: Outcomes Assessor
Masking Description: An independent assessor who is blinded to the group allocations will assess the participants' outcomes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- BCE Combination group (Experimental): 16-week BCE programme with exercise training.
  Six 1-hour sessions of BCE programme and a weekly 45-60 minute centre-based exercise programme from week 4 to week 16.
  Interventions: Other: BCE Combination group
- Exercise group (No Intervention): 16-week programme with health talks and exercise training.
  Six 1-hour sessions of health talks and a weekly 45-60 minutes centre-based exercise programme from week 4 to week 16.
- Control group (No Intervention): Six sessions of centre-based health talks on the management of different health issues with the exception of fatigue.

INTERVENTIONS:
Other: BCE Combination group — The combination intervention programme consists of a weekly exercise training sessions and 6 sessions of Behavioral Change Enhancement (BCE) programme.
  Arms: BCE Combination group

SUMMARY:
This project aims to investigate the effects of an individualized exercise programme with and without BCE strategies for community-dwelling frail older people with general fatigue, so as to reduce their fatigue and improve their physical endurance, exercise self-efficacy, and habitual physical activity, while reducing their symptoms of frailty.

Twelve district community health centres will be randomized to one of the three study groups: the combined (COMB) group, receiving the 16-week combined intervention consisting of individualized exercise training and Behavioural Change Enhancement programmes plus two booster sessions at 2 and 6 months after the programme; the exercise (EXER) group, receiving exercise training and health talks only; or the control group, receiving health talks only. Participants from each centre will be placed in their centre's corresponding group.

It is hypothesized that the COMB group will achieve a significantly greater reduction in fatigue and a greater improvement in their physical endurance, exercise self-efficacy, and habitual physical activity, and a significantly greater reduction in their frailty symptoms, when compared with the EXER and control groups at 1 week and 6 and 12 months after completing the interventions.

DETAILED DESCRIPTION:
All twelve community centres, which provide similar types of community care and social support services for community-dwelling older people, have been invited by a convenience method to work as collaborators in this study. The target population of this study are community-dwelling frail older people with general fatigue with a nonspecific cause who will be recruited through the community centres. Using computer-generated random numbers, a biostatistician not affiliated with this study will randomize the centres into either: control, EXER, or COMB. The number of participants recruited in each centre will be in proportion to the size of the centre.

Participants allocated to the COMB group will receive a 16-week programme with a combination of the BCE programme and exercise training. The BCE programme is designed based on the Health Action Process Approach (HAPA) model and was piloted by the principal investigator, which aims to motivate the participants to develop the intention to actively manage their fatigue; and to encourage them to gradually exceed the perceived limits of their energy and to recondition their bodies by participating in exercise according to their individual exercise regimens. The BCE programme consists of three phases (the goal initiation, plan formulation and action execution) with 6 face-to-face 1-hour sessions plus two booster BCE sessions at 2 and 6 months after the programme.

For the exercise training, a weekly 45-60 minute centre-based exercise programme, which is designed according to the American Heart Association's recommendations on exercise for older people will be arranged from weeks 4-16 during the execution phase. The exercise sessions consist of balance training, resistance exercises, and aerobic training. All participants will receive circuit training with set exercises, but the dosage of different components will be tailor-made for each participant by a physiotherapist after having their physical conditions examined.

The EXER group will receive a 16-week programme with a combination of exercise training and centre-based health talks on the management of different health issues with the exception of fatigue.

The control group will attend centre-based health talks only.

The number and timing of the health talks for the other two groups will be similar to those in the BCE sessions.

ELIGIBILITY:
Inclusion Criteria:

* community-dwelling older people aged > 70 years;
* able to communicate in Cantonese to ensure that they understand our instructions;
* able to walk with or without an assistive device and able to complete the Time Up and Go (TUG) test with no specific cutoff point to ensure that their mobility and balance is good enough to join the exercise training; and
* in a frail state with exhaustion as determined using the Fried Frailty Index (FFI), including: i) an unintentional loss of 10% of body weight in the past year; ii) exhaustion: by answering 'Yes' to either 'I felt that everything I did was an effort', or 'I could not get going in the last week'; iii) a slow walk time: with an average walking speed in the lowest quintile stratified by median body height; iv) reduced grip strength: with maximal grip strength in the lowest quintile stratified by body mass index quartile; and v) the Physical Activity Scale for the Elderly-Chinese (PASE-C) score in the lowest quintile (i.e., < 30 for men and < 27.7 for women). The presence of > 3 items indicates frailty, and one criterion indicates that they suffer from exhaustion.

Exclusion Criteria: are older people who:

* are suffering from any disease in which fatigue is a dominant symptom (such as neurodegenerative diseases, cancer, and end-stage renal failure cachexia cases;
* have been hospitalized for > 5 days in the preceding 3 months, which may lead to muscle wasting due to recent bed rest or reduced activity levels during hospitalization;
* underwent major surgery (such as total joint replacement, major abdominal surgeries) during the last 6 months;
* are confined to bed or restricted by the permanent use of a wheelchair;
* report that they regularly perform moderately intense exercise (such as hiking, Tai Chi) for > 3 hours per week;
* are terminally ill;
* have been diagnosed with major depression entailing frequent adjustments of their antidepressants to control unstable depressive moods. The criteria were chosen to avoid recruiting people with depression-induced fatigue. However, a consistent feeling of fatigue may manifest as a depressed mood. Thus, the participants' mood will be assessed using the Chinese-Geriatric Depression Scale (C-GDS).

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 184 (Actual)
Dates: Start 2018-02-26 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2021-01-01 (Actual)

PRIMARY OUTCOMES:
Participants' level of fatigue will be assessed using the 20-item Chinese Multidimensional Fatigue Inventory (CMFI-20) | To detect the change from baseline total fatigue score at mid-term programme (i.e. wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after completing the programme
  CMFI-20 consists of 20 items, each item is rated on a 5-point Likert scale from 1=strongly agree to 5 = strongly disagree, with all items summed to get the total score which ranges from 20-100, a higher score indicates more fatigue.

SECONDARY OUTCOMES:
Participants' lower-limb strength will be assessed using the 30-second chair stand test | To detect the change from baseline lower-limb strength at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after completing the programme
  Participants will be asked to stand up and sit down as many as they can within 30 seconds on a standard chair. The total number of standing up from a chair will be counted. More number indicates better lower-limb strength
Participants' upper-limb strength will be assessed using a handheld Jamar Hydraulic Hand Dynamometer | To detect the change from baseline upper-limb strength in kg at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after completing the programme
  It will be measured by handheld Jamar Hydraulic Hand Dynamometer with kilogram (kg). Greater force in kg indicates better upper-limb strength
Participants' functional mobility will be measured by the timed-up-and-go-test | To detect the change from baseline time to complete the "timed-up-and-go-test" at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after completing the programme
  Record the time in second that participants complete the timed up and go test to indicate their functional mobility
Participants' gait speed will be measured by the 6 meter walk test | To detect the change from baseline gait speed at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after the completion of the programme
  Record the time in second that participants complete the 6 meter walk test to indicate the their gait speed.
Participants' exercise self-efficacy will be measured using Chinese Self-Efficacy for Exercise (CSEE) scale | To detect the change from baseline total CSSE score at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after completing the programme
  The CSEE scale contains of 9 items. Each item is rated on 11-point Liker scale from 0 = no confidence to 10 = full of confidence. All item scores are summed to get the total score which ranges from 0 to 90 with a higher score indicates higher exercise self-efficacy
Participants' frailty level will be assessed using Fried Frailty Index (FFI) | To detect the change from baseline frailty level at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after the completion of the programme
  Fried Frailty Index includes: i) an unintentional loss of 10% of body weight in the past year; ii) exhaustion: by answering 'Yes' to either 'I felt that everything I did was an effort', or 'I could not get going in the last week'; iii) a slow walk time: with an average walking speed in the lowest quintile stratified by median body height; iv) reduced handgrip strength: with maximal grip strength in the lowest quintile stratified by body mass index quartile; and v) the Physical Activity Scale for the Elderly-Chinese (PASE-C) score in the lowest quintile (i.e., < 30 for men and < 27.7 for women).
Physical activity will be assessed using the Physical Activity Scale for the Elderly-Chinese (PASE-C) | To detect the change from baseline PASE-C total score at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after completing the programme
  The PASE-C is a self-reported scale for evaluating the level of physical activity of older people over a 1-week period. It consists of 12-items to explain three levels of activities: leisure time activity, household activity and work-related activity. Basic descriptions are:1) 5-items under the leisure time activity are rated on a 4-point scale; 2) 6-items relate to household activity are rated on dichotomous (yes or no) scale; 3) work-related activity is rated by whether the activity is a paid or volunteer work; 4) The duration (in hours) spent on such activities will be reported by the participants. 5) The total PASE-C score will be calculated by adding the score of each item determined on the basis of the time spent on each activity or the presence or absence of activity over the past 7 days.6) Amount of time spent in each activity multiplied by PASE-C item weights & adding all scores together for the final PASE-C score. A high score indicates a high level of physical activity.
Participants' depressive mood will be assessed by the 15-item Chinese version Geriatric Depression Scale (C-GDS) | To detect the change from baseline C-GDS total score at mid-term programme (wk 8 after commences of the programme),and then 1 week, 6 month and 12 months months after the completion of the programme
  The C-GDS consists of 15 yes/no questions. Each negative answer will be given 1 point, with possible scores ranging from 0-15. The higher score indicates more depressive mood. • Respondents with a score more than 8 are identified as having symptoms of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Yat-wa Justina Liu, Principal Investigator — The Hong Kong Polytechnic University
Locations (1):
- Justina Liu, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
For confidentiality, the data will be kept anonymous and the names of all participants will be replaced by reference codes. The data collected will be kept in a locked place and electronic versions will be encrypted, and only be accessible by the researchers. All data will be destroyed within 3 years after the completion of this research.

REFERENCES:
- [Background] Avlund K. Fatigue in older adults: an early indicator of the aging process? Aging Clin Exp Res. 2010 Apr;22(2):100-15. doi: 10.1007/BF03324782. PMID 20440097
- [Background] Xue QL, Bandeen-Roche K, Varadhan R, Zhou J, Fried LP. Initial manifestations of frailty criteria and the development of frailty phenotype in the Women's Health and Aging Study II. J Gerontol A Biol Sci Med Sci. 2008 Sep;63(9):984-90. doi: 10.1093/gerona/63.9.984. PMID 18840805
- [Background] Gill TM, Desai MM, Gahbauer EA, Holford TR, Williams CS. Restricted activity among community-living older persons: incidence, precipitants, and health care utilization. Ann Intern Med. 2001 Sep 4;135(5):313-21. doi: 10.7326/0003-4819-135-5-200109040-00007. PMID 11529694
- [Background] Schultz-Larsen K, Avlund K. Tiredness in daily activities: a subjective measure for the identification of frailty among non-disabled community-living older adults. Arch Gerontol Geriatr. 2007 Jan-Feb;44(1):83-93. doi: 10.1016/j.archger.2006.03.005. Epub 2006 Nov 13. PMID 17095107
- [Background] Hardy SE, Studenski SA. Fatigue and function over 3 years among older adults. J Gerontol A Biol Sci Med Sci. 2008 Dec;63(12):1389-92. doi: 10.1093/gerona/63.12.1389. PMID 19126853
- [Background] Avlund K, Damsgaard MT, Schroll M. Tiredness as determinant of subsequent use of health and social services among nondisabled elderly people. J Aging Health. 2001 May;13(2):267-86. doi: 10.1177/089826430101300206. PMID 11787515
- [Background] Fried LP, Tangen CM, Walston J, Newman AB, Hirsch C, Gottdiener J, Seeman T, Tracy R, Kop WJ, Burke G, McBurnie MA; Cardiovascular Health Study Collaborative Research Group. Frailty in older adults: evidence for a phenotype. J Gerontol A Biol Sci Med Sci. 2001 Mar;56(3):M146-56. doi: 10.1093/gerona/56.3.m146. PMID 11253156
- [Background] Drey M, Pfeifer K, Sieber CC, Bauer JM. The Fried frailty criteria as inclusion criteria for a randomized controlled trial: personal experience and literature review. Gerontology. 2011;57(1):11-8. doi: 10.1159/000313433. Epub 2010 Apr 21. PMID 20407227
- [Background] Moschny A, Platen P, Klaassen-Mielke R, Trampisch U, Hinrichs T. Barriers to physical activity in older adults in Germany: a cross-sectional study. Int J Behav Nutr Phys Act. 2011 Nov 2;8:121. doi: 10.1186/1479-5868-8-121. PMID 22047024
- [Background] Rasinaho M, Hirvensalo M, Leinonen R, Lintunen T, Rantanen T. Motives for and barriers to physical activity among older adults with mobility limitations. J Aging Phys Act. 2007 Jan;15(1):90-102. doi: 10.1123/japa.15.1.90. PMID 17387231
- [Background] Clark LV, White PD. The role of deconditioning and therapeutic exercise in chronic fatigue syndrome (CFS). Journal of Mental Health. 2005; 14(3): 237-52.
- [Background] Yu DS, Lee DT, Man NW. Fatigue among older people: a review of the research literature. Int J Nurs Stud. 2010 Feb;47(2):216-28. doi: 10.1016/j.ijnurstu.2009.05.009. Epub 2009 Jun 12. PMID 19524240
- [Background] Smets EM, Garssen B, Bonke B, De Haes JC. The Multidimensional Fatigue Inventory (MFI) psychometric qualities of an instrument to assess fatigue. J Psychosom Res. 1995 Apr;39(3):315-25. doi: 10.1016/0022-3999(94)00125-o. PMID 7636775
- [Background] Liu JY, Lai CK, Siu PM, Kwong E, Tse MM. An individualized exercise programme with and without behavioural change enhancement strategies for managing fatigue among frail older people: a quasi-experimental pilot study. Clin Rehabil. 2017 Apr;31(4):521-531. doi: 10.1177/0269215516649226. Epub 2016 Jul 10. PMID 27162189
- [Background] Egerton T. Self-reported aging-related fatigue: a concept description and its relevance to physical therapist practice. Phys Ther. 2013 Oct;93(10):1403-13. doi: 10.2522/ptj.20130011. Epub 2013 May 23. PMID 23704037
- [Background] Hellstrom Y, Persson G, Hallberg IR. Quality of life and symptoms among older people living at home. J Adv Nurs. 2004 Dec;48(6):584-93. doi: 10.1111/j.1365-2648.2004.03247.x. PMID 15548249
- [Background] Ream E, Richardson A. Fatigue: a concept analysis. Int J Nurs Stud. 1996 Oct;33(5):519-29. doi: 10.1016/0020-7489(96)00004-1. PMID 8886902
- [Background] Avlund K, Pedersen AN, Schroll M. Functional decline from age 80 to 85: influence of preceding changes in tiredness in daily activities. Psychosom Med. 2003 Sep-Oct;65(5):771-7. doi: 10.1097/01.psy.0000082640.61645.bf. PMID 14508019
- [Background] Fried LP, Ferrucci L, Darer J, Williamson JD, Anderson G. Untangling the concepts of disability, frailty, and comorbidity: implications for improved targeting and care. J Gerontol A Biol Sci Med Sci. 2004 Mar;59(3):255-63. doi: 10.1093/gerona/59.3.m255. PMID 15031310
- [Background] Santos-Eggimann B, Cuenoud P, Spagnoli J, Junod J. Prevalence of frailty in middle-aged and older community-dwelling Europeans living in 10 countries. J Gerontol A Biol Sci Med Sci. 2009 Jun;64(6):675-81. doi: 10.1093/gerona/glp012. Epub 2009 Mar 10. PMID 19276189
- [Background] Ble A, Cherubini A, Volpato S, Bartali B, Walston JD, Windham BG, Bandinelli S, Lauretani F, Guralnik JM, Ferrucci L. Lower plasma vitamin E levels are associated with the frailty syndrome: the InCHIANTI study. J Gerontol A Biol Sci Med Sci. 2006 Mar;61(3):278-83. doi: 10.1093/gerona/61.3.278. PMID 16567378
- [Background] Cramp F, Daniel J. Exercise for the management of cancer-related fatigue in adults. Cochrane Database Syst Rev. 2008 Apr 16;(2):CD006145. doi: 10.1002/14651858.CD006145.pub2. PMID 18425939
- [Background] Neill J, Belan I, Ried K. Effectiveness of non-pharmacological interventions for fatigue in adults with multiple sclerosis, rheumatoid arthritis, or systemic lupus erythematosus: a systematic review. J Adv Nurs. 2006 Dec;56(6):617-35. doi: 10.1111/j.1365-2648.2006.04054.x. PMID 17118041
- [Background] Martin KA, Sinden AR. Who will stay and who will go? A review of older adults' adherence to randomized controlled trials of exercise. J Aging Phys Act. 2001; 9(2): 91-114.
- [Background] Larun L, Brurberg KG, Odgaard-Jensen J, Price JR. Exercise therapy for chronic fatigue syndrome. status and date: New search for studies and content updated (no change to conclusions), published in. 2015; (2).
- [Background] Edmonds M, McGuire H, Price J. Exercise therapy for chronic fatigue syndrome. Cochrane Database Syst Rev. 2004;(3):CD003200. doi: 10.1002/14651858.CD003200.pub2. PMID 15266475
- [Background] Jones DE, Gray JC, Newton J. Perceived fatigue is comparable between different disease groups. QJM. 2009 Sep;102(9):617-24. doi: 10.1093/qjmed/hcp091. Epub 2009 Jul 24. PMID 19633030
- [Background] Liu CJ, Latham NK. Progressive resistance strength training for improving physical function in older adults. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD002759. doi: 10.1002/14651858.CD002759.pub2. PMID 19588334
- [Background] Clegg AP, Barber SE, Young JB, Forster A, Iliffe SJ. Do home-based exercise interventions improve outcomes for frail older people? Findings from a systematic review. Rev Clin Gerontol. 2012 Feb;22(1):68-78. doi: 10.1017/S0959259811000165. Epub 2012 Aug 24. PMID 27226701
- [Background] Simons R, Andel R. The effects of resistance training and walking on functional fitness in advanced old age. J Aging Health. 2006 Feb;18(1):91-105. doi: 10.1177/0898264305281102. PMID 16470977
- [Background] Network NCC. NCCN clinical practice guideline in oncology: cancer-related fatigue. Available from: www nccn org. 2013.
- [Background] Theou O, Stathokostas L, Roland KP, Jakobi JM, Patterson C, Vandervoort AA, Jones GR. The effectiveness of exercise interventions for the management of frailty: a systematic review. J Aging Res. 2011 Apr 4;2011:569194. doi: 10.4061/2011/569194. PMID 21584244
- [Background] Pinto BM, Frierson GM, Rabin C, Trunzo JJ, Marcus BH. Home-based physical activity intervention for breast cancer patients. J Clin Oncol. 2005 May 20;23(15):3577-87. doi: 10.1200/JCO.2005.03.080. PMID 15908668
- [Background] Schwarzer R. Modeling health behavior change: How to predict and modify the adoption and maintenance of health behaviors. Appl Psychol-Int Rev. 2008; 57(1): 1 - 29.
- [Background] Lippke S, Ziegelmann JP, Schwarzer R. Behavioral intentions and action plans promote physical exercise: a longitudinal study with orthopedic rehabilitation patients. J Sport Exerc Psychol. 2004; 26(3): 470.
- [Background] Scholz U, Sniehotta FF, Burkert S, Schwarzer R. Increasing physical exercise levels: age-specific benefits of planning. J Aging Health. 2007 Oct;19(5):851-66. doi: 10.1177/0898264307305207. PMID 17827449
- [Background] Ghisi GL, Grace SL, Thomas S, Oh P. Behavior determinants among cardiac rehabilitation patients receiving educational interventions: an application of the health action process approach. Patient Educ Couns. 2015 May;98(5):612-21. doi: 10.1016/j.pec.2015.01.006. Epub 2015 Jan 20. PMID 25638305
- [Background] Evers A, Klusmann V, Schwarzer R, Heuser I. Adherence to physical and mental activity interventions: coping plans as a mediator and prior adherence as a moderator. Br J Health Psychol. 2012 Sep;17(3):477-91. doi: 10.1111/j.2044-8287.2011.02049.x. Epub 2011 Sep 5. PMID 22107076
- [Background] Chien WT, Bressington D. A randomized controlled clinical trial of a nurse-led structured psychosocial intervention program for people with first-onset mental illness in psychiatric outpatient clinics. Psychiatry Res. 2015 Sep 30;229(1-2):277-86. doi: 10.1016/j.psychres.2015.07.012. Epub 2015 Jul 10. PMID 26193827
- [Background] Chien WT, Mui JH, Cheung EF, Gray R. Effects of motivational interviewing-based adherence therapy for schizophrenia spectrum disorders: a randomized controlled trial. Trials. 2015 Jun 14;16:270. doi: 10.1186/s13063-015-0785-z. PMID 26072311
- [Background] Tan PJ, Khoo EM, Chinna K, Hill KD, Poi PJ, Tan MP. An individually-tailored multifactorial intervention program for older fallers in a middle-income developing country: Malaysian Falls Assessment and Intervention Trial (MyFAIT). BMC Geriatr. 2014 Jun 21;14:78. doi: 10.1186/1471-2318-14-78. PMID 24951180
- [Background] Craig P, Dieppe P, Macintyre S, Michie S, Nazareth I, Petticrew M; Medical Research Council Guidance. Developing and evaluating complex interventions: the new Medical Research Council guidance. BMJ. 2008 Sep 29;337:a1655. doi: 10.1136/bmj.a1655. PMID 18824488
- [Background] Hemming K, Girling AJ, Sitch AJ, Marsh J, Lilford RJ. Sample size calculations for cluster randomised controlled trials with a fixed number of clusters. BMC Med Res Methodol. 2011 Jun 30;11:102. doi: 10.1186/1471-2288-11-102. PMID 21718530
- [Background] Wijeratne C, Hickie I, Brodaty H. The characteristics of fatigue in an older primary care sample. J Psychosom Res. 2007 Feb;62(2):153-8. doi: 10.1016/j.jpsychores.2006.09.011. PMID 17270573
- [Background] Woo J, Ho SC, Lau J, Yuen YK, Chiu H, Lee HC, Chi I. The prevalence of depressive symptoms and predisposing factors in an elderly Chinese population. Acta Psychiatr Scand. 1994 Jan;89(1):8-13. doi: 10.1111/j.1600-0447.1994.tb01478.x. PMID 8140912
- [Background] Lee LL, Arthur A, Avis M. Using self-efficacy theory to develop interventions that help older people overcome psychological barriers to physical activity: a discussion paper. Int J Nurs Stud. 2008 Nov;45(11):1690-9. doi: 10.1016/j.ijnurstu.2008.02.012. Epub 2008 May 22. PMID 18501359
- [Background] Hinrichs T, Moschny A, Brach M, Wilm S, Klaassen-Mielke R, Trampisch M, Platen P. Effects of an exercise programme for chronically ill and mobility-restricted elderly with structured support by the general practitioner's practice (HOMEfit) - study protocol of a randomised controlled trial. Trials. 2011 Dec 21;12:263. doi: 10.1186/1745-6215-12-263. PMID 22188781
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C; American College of Sports Medicine; American Heart Association. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Circulation. 2007 Aug 28;116(9):1094-105. doi: 10.1161/CIRCULATIONAHA.107.185650. Epub 2007 Aug 1. PMID 17671236
- [Background] Chin A Paw MJ, de Jong N, Schouten EG, Hiddink GJ, Kok FJ. Physical exercise and/or enriched foods for functional improvement in frail, independently living elderly: a randomized controlled trial. Arch Phys Med Rehabil. 2001 Jun;82(6):811-7. doi: 10.1053/apmr.2001.23278. PMID 11387588
- [Background] Charlson ME, Pompei P, Ales KL, MacKenzie CR. A new method of classifying prognostic comorbidity in longitudinal studies: development and validation. J Chronic Dis. 1987;40(5):373-83. doi: 10.1016/0021-9681(87)90171-8. PMID 3558716
- [Background] Tian J, Hong JS. Validation of the Chinese version of Multidimensional Fatigue Inventory-20 in Chinese patients with cancer. Support Care Cancer. 2012 Oct;20(10):2379-83. doi: 10.1007/s00520-011-1357-8. Epub 2011 Dec 24. PMID 22198167
- [Background] Rikli R, Jones C. Development and validation of a functional fitness test for community-residing older adults. J Aging Phys Act. 1999; 7(2): 129 - 61.
- [Background] Yang XJ, Hill K, Moore K, Williams S, Dowson L, Borschmann K, Simpson JA, Dharmage SC. Effectiveness of a targeted exercise intervention in reversing older people's mild balance dysfunction: a randomized controlled trial. Phys Ther. 2012 Jan;92(1):24-37. doi: 10.2522/ptj.20100289. Epub 2011 Oct 6. PMID 21979272
- [Background] Resnick B, Jenkins LS. Testing the reliability and validity of the Self-Efficacy for Exercise scale. Nurs Res. 2000 May-Jun;49(3):154-9. doi: 10.1097/00006199-200005000-00007. PMID 10882320
- [Background] Washburn RA, Smith KW, Jette AM, Janney CA. The Physical Activity Scale for the Elderly (PASE): development and evaluation. J Clin Epidemiol. 1993 Feb;46(2):153-62. doi: 10.1016/0895-4356(93)90053-4. PMID 8437031
- [Background] Ku P-W, Sun W-J, Chang C-Y, Chen L-J. Reliability and validity of the Chinese version of the Physical Activity Scale for the Elderly. Sports & Exercise Research. 2013; 15(3): 309-19.
- [Background] Ngai SP, Cheung RT, Lam PL, Chiu JK, Fung EY. Validation and reliability of the Physical Activity Scale for the Elderly in Chinese population. J Rehabil Med. 2012 May;44(5):462-5. doi: 10.2340/16501977-0953. PMID 22549657
- [Background] Chan AC. Clinical validation of the Geriatric Depression Scale (GDS): Chinese version. J Aging Health. 1996 May;8(2):238-53. doi: 10.1177/089826439600800205. PMID 10160560
- [Background] Bellg AJ, Borrelli B, Resnick B, Hecht J, Minicucci DS, Ory M, Ogedegbe G, Orwig D, Ernst D, Czajkowski S; Treatment Fidelity Workgroup of the NIH Behavior Change Consortium. Enhancing treatment fidelity in health behavior change studies: best practices and recommendations from the NIH Behavior Change Consortium. Health Psychol. 2004 Sep;23(5):443-51. doi: 10.1037/0278-6133.23.5.443. PMID 15367063
- [Background] Stevens JP. Applied multivariate statistics for the social sciences: Routledge; 2012.
- [Background] Krippendorff K. Content analysis: An introduction to its methodology: Sage; 2004.
- [Derived] Liu JYW, Yin YH, Kor PPK, Kwan RYC, Lee PH, Chien WT, Siu PM, Hill KD. Effects of an individualised exercise programme plus Behavioural Change Enhancement (BCE) strategies for managing fatigue in frail older adults: a cluster randomised controlled trial. BMC Geriatr. 2023 Jun 16;23(1):370. doi: 10.1186/s12877-023-04080-0. PMID 37328797
- [Derived] Liu JYW, Kor PPK, Lee PL, Chien WT, Siu PM, Hill KD. Effects of an Individualized Exercise Program Plus Behavioral Change Enhancement Strategies for Managing Fatigue in Older People Who Are Frail: Protocol for a Cluster Randomized Controlled Trial. Phys Ther. 2019 Dec 16;99(12):1616-1627. doi: 10.1093/ptj/pzz130. PMID 31508798

DOCUMENTS (3):
  • Study Protocol (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03394495/Prot_001.pdf
  • Statistical Analysis Plan (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03394495/SAP_002.pdf
  • Informed Consent Form (2017-12-15): https://cdn.clinicaltrials.gov/large-docs/95/NCT03394495/ICF_000.pdf